CLINICAL TRIAL: NCT01006980
Title: BRIM 3: A Randomized, Open-Label, Controlled, Multicenter, Phase III Study in Previously Untreated Patients With Unresectable Stage IIIC or Stage IV Melanoma With V600E BRAF Mutation Receiving Vemurafenib (RO5185426) or Dacarbazine
Brief Title: A Study of Vemurafenib (RO5185426) in Comparison With Dacarbazine in Previously Untreated Patients With Metastatic Melanoma (BRIM 3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO25026; 2009-012293-12
Record Dates: First submitted 2009-10-30; First posted 2009-11-03 (Estimated); Results first posted 2011-11-16 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2015-12

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib; Dacarbazine

ARMS (2):
- Vemurafenib (Experimental)
  Interventions: Drug: Vemurafenib
- Dacarbazine (Active Comparator)
  Interventions: Drug: Dacarbazine

INTERVENTIONS:
Drug: Vemurafenib — 960 mg (as 240 mg tables) orally twice daily
  Other Names: Zelboraf®; RO5185426
  Arms: Vemurafenib
Drug: Dacarbazine — 1000 mg/m2 intravenously every 3 weeks
  Arms: Dacarbazine

SUMMARY:
This randomized, open-label study evaluated the efficacy, safety and tolerability of vemurafenib (RO5185426) as compared to dacarbazine in previously untreated patients with metastatic melanoma. Patients were randomized to receive either vemurafenib 960 mg orally twice daily or dacarbazine 1000 mg/m2 intravenously every 3 weeks. Study treatment was continued until disease progression or unacceptable toxicity occurred. The data and safety monitoring board recommended that patients in the dacarbazine group be allowed to cross over to receive vemurafenib, and the protocol was amended accordingly on January 14, 2011, as both overall survival and progression-free survival endpoints had met the prespecified criteria for statistical significance in favor of vemurafenib.

ELIGIBILITY:
Inclusion Criteria:

* adults, >/=18 years of age
* metastatic melanoma, stage IIIC or IV (AJCC)
* treatment-naïve (no prior systemic anticancer therapy)
* positive for BRAF V600E mutation
* measurable disease by RECIST criteria
* negative pregnancy test and, for fertile men and women, effective contraception during treatment and for 6 months after completion

Exclusion Criteria:

* active central nervous system metastases
* history of carcinomatous meningitis
* severe cardiovascular disease within 6 months prior to study drug administration
* previous malignancy within 5 years prior to study, except for basal or squamous cell carcinoma of the skin, melanoma in-situ, or carcinoma in-situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 675 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (98):
- United States (20):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Los Angeles, California
  - San Francisco, California
  - Santa Monica, California
  - Aurora, Colorado
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - Detroit, Michigan
  - St Louis, Missouri
  - New York, New York
  - Chapel Hill, North Carolina
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
- Australia (10):
  - Brisbane
  - Frankston
  - Malvern
  - Melbourne
  - Nedlands
  - Newcastle
  - St Leonards
  - Sydney
  - Westmead
  - Woolloongabba
- Canada (6):
  - Edmonton, Alberta
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- France (10):
  - Bordeaux
  - Lille
  - Marseille
  - Montpellier
  - Nantes
  - Nice
  - Paris
  - Pierre-Bénite
  - Rouen
  - Villejuif
- Germany (17):
  - Buxtehude
  - Cologne
  - Dresden
  - Erfurt
  - Essen
  - Frankfurt
  - Hanover
  - Heidelberg
  - Jena
  - Kiel
  - Leipzig
  - Mainz
  - Minden
  - München
  - Regensburg
  - Tübingen
  - Würzburg
- Israel (3):
  - Jerusalem
  - Ramat Gan
  - Tel Aviv
- Italy (6):
  - Bari
  - Genova
  - Milan
  - Napoli
  - Roma
  - Siena
- Netherlands (2):
  - Amsterdam
  - Groningen
- New Zealand (5):
  - Auckland
  - Dunedin
  - Hamilton
  - Palmerston North
  - Wellington
- Sweden (5):
  - Linköping
  - Lund
  - Stockholm
  - Umeå
  - Uppsala
- Switzerland (2):
  - Lausanne
  - Zurich
- United Kingdom (12):
  - Cambridge
  - Edinburgh
  - Glasgow
  - London
  - Manchester
  - Newcastle upon Tyne
  - Northwood
  - Nottingham
  - Oxford
  - Southampton
  - Sutton
  - Swansea

REFERENCES:
- [Derived] Ascierto PA, Ribas A, Larkin J, McArthur GA, Lewis KD, Hauschild A, Flaherty KT, McKenna E, Zhu Q, Mun Y, Dreno B. Impact of initial treatment and prognostic factors on postprogression survival in BRAF-mutated metastatic melanoma treated with dacarbazine or vemurafenib +/- cobimetinib: a pooled analysis of four clinical trials. J Transl Med. 2020 Aug 3;18(1):294. doi: 10.1186/s12967-020-02458-x. PMID 32746839
- [Derived] Chapman PB, Robert C, Larkin J, Haanen JB, Ribas A, Hogg D, Hamid O, Ascierto PA, Testori A, Lorigan PC, Dummer R, Sosman JA, Flaherty KT, Chang I, Coleman S, Caro I, Hauschild A, McArthur GA. Vemurafenib in patients with BRAFV600 mutation-positive metastatic melanoma: final overall survival results of the randomized BRIM-3 study. Ann Oncol. 2017 Oct 1;28(10):2581-2587. doi: 10.1093/annonc/mdx339. PMID 28961848
- [Derived] Yamazaki N, Kiyohara Y, Sugaya N, Uhara H. Phase I/II study of vemurafenib in patients with unresectable or recurrent melanoma with BRAF(V) (600) mutations. J Dermatol. 2015 Jul;42(7):661-6. doi: 10.1111/1346-8138.12873. Epub 2015 Apr 17. PMID 25884515
- [Derived] Frederick DT, Salas Fragomeni RA, Schalck A, Ferreiro-Neira I, Hoff T, Cooper ZA, Haq R, Panka DJ, Kwong LN, Davies MA, Cusack JC, Flaherty KT, Fisher DE, Mier JW, Wargo JA, Sullivan RJ. Clinical profiling of BCL-2 family members in the setting of BRAF inhibition offers a rationale for targeting de novo resistance using BH3 mimetics. PLoS One. 2014 Jul 1;9(7):e101286. doi: 10.1371/journal.pone.0101286. eCollection 2014. PMID 24983357
- [Derived] McArthur GA, Chapman PB, Robert C, Larkin J, Haanen JB, Dummer R, Ribas A, Hogg D, Hamid O, Ascierto PA, Garbe C, Testori A, Maio M, Lorigan P, Lebbe C, Jouary T, Schadendorf D, O'Day SJ, Kirkwood JM, Eggermont AM, Dreno B, Sosman JA, Flaherty KT, Yin M, Caro I, Cheng S, Trunzer K, Hauschild A. Safety and efficacy of vemurafenib in BRAF(V600E) and BRAF(V600K) mutation-positive melanoma (BRIM-3): extended follow-up of a phase 3, randomised, open-label study. Lancet Oncol. 2014 Mar;15(3):323-32. doi: 10.1016/S1470-2045(14)70012-9. Epub 2014 Feb 7. PMID 24508103
- [Derived] Lacouture ME, Duvic M, Hauschild A, Prieto VG, Robert C, Schadendorf D, Kim CC, McCormack CJ, Myskowski PL, Spleiss O, Trunzer K, Su F, Nelson B, Nolop KB, Grippo JF, Lee RJ, Klimek MJ, Troy JL, Joe AK. Analysis of dermatologic events in vemurafenib-treated patients with melanoma. Oncologist. 2013;18(3):314-22. doi: 10.1634/theoncologist.2012-0333. Epub 2013 Mar 1. PMID 23457002
- [Derived] Su F, Viros A, Milagre C, Trunzer K, Bollag G, Spleiss O, Reis-Filho JS, Kong X, Koya RC, Flaherty KT, Chapman PB, Kim MJ, Hayward R, Martin M, Yang H, Wang Q, Hilton H, Hang JS, Noe J, Lambros M, Geyer F, Dhomen N, Niculescu-Duvaz I, Zambon A, Niculescu-Duvaz D, Preece N, Robert L, Otte NJ, Mok S, Kee D, Ma Y, Zhang C, Habets G, Burton EA, Wong B, Nguyen H, Kockx M, Andries L, Lestini B, Nolop KB, Lee RJ, Joe AK, Troy JL, Gonzalez R, Hutson TE, Puzanov I, Chmielowski B, Springer CJ, McArthur GA, Sosman JA, Lo RS, Ribas A, Marais R. RAS mutations in cutaneous squamous-cell carcinomas in patients treated with BRAF inhibitors. N Engl J Med. 2012 Jan 19;366(3):207-15. doi: 10.1056/NEJMoa1105358. PMID 22256804
- [Derived] Chapman PB, Hauschild A, Robert C, Haanen JB, Ascierto P, Larkin J, Dummer R, Garbe C, Testori A, Maio M, Hogg D, Lorigan P, Lebbe C, Jouary T, Schadendorf D, Ribas A, O'Day SJ, Sosman JA, Kirkwood JM, Eggermont AM, Dreno B, Nolop K, Li J, Nelson B, Hou J, Lee RJ, Flaherty KT, McArthur GA; BRIM-3 Study Group. Improved survival with vemurafenib in melanoma with BRAF V600E mutation. N Engl J Med. 2011 Jun 30;364(26):2507-16. doi: 10.1056/NEJMoa1103782. Epub 2011 Jun 5. PMID 21639808

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 675 participants were randomized, 337 to vemurafenib and 338 to dacarbazine. One participant randomized to dacarbazine was treated in error with vemurafenib throughout the study and is included in the Vemurafenib arm in the table below and for exposure and safety analyses and is included in the dacarbazine arm for efficacy analyses.
Groups:
- Vemurafenib: Participants received continuous oral doses of vemurafenib (RO5185426) 960 mg twice a day. Participants took four 240 mg tablets in the morning and four 240 mg tablets in the evening (960 mg twice a day for a total daily dose of 1920 mg).
- Dacarbazine: Dacarbazine was administered intravenously 1000 mg/m˄2 up to 60 minutes on Day 1 of every 3 weeks (3 weeks was one cycle length).
Period: Vemurafenib and Dacarbazine
Arm/Group | Vemurafenib | Dacarbazine
Started | 337 | 338
Treated | 336 | 293
Completed | 0 | 0
Not Completed | 337 | 338
Not completed — Randomized but Not Treated | 1 | 45
Not completed — Adverse Event | 25 | 5
Not completed — Death | 13 | 12
Not completed — Progression | 257 | 218
Not completed — Withdrawal of Consent | 4 | 6
Not completed — Refuse Treatment | 9 | 6
Not completed — Protocol Violation | 2 | 3
Not completed — Reason Not Specified | 26 | 43
Period: Crossover: Dacarbazine to Vemurafenib
Arm/Group | Vemurafenib | Dacarbazine
Started | 0 | 84 (Participants who crossed over from dacarbazine to vemurafenib treatment.)
Completed | 0 | 0
Not Completed | 0 | 84
Not completed — Adverse Event | 0 | 4
Not completed — Death | 0 | 4
Not completed — Progression | 0 | 65
Not completed — Withdrawal of Consent | 0 | 1
Not completed — Reason Not Specified | 0 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vemurafenib | Dacarbazine | Total
Number analyzed (Participants) | 337 | 338 | 675
Age, Customized [Number; unit: participants]
  < 65 years | 244 | 270 | 514
  >=65 years | 93 | 68 | 161
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 157 | 294
  Male | 200 | 181 | 381

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: An Overall survival event was defined as death due to any cause. The number of participants with overall survival events is reported.
Time Frame: From randomization (initiated January 2010) to December 30 2010. Median follow-up time in the vemurafenib group was 3.75 months (range 0.3 to 10.8) and in the dacarbazine group was 2.33 months (range <0.1 to 10.3).
Population: The intent-to-treat (ITT) population was defined as all randomized participants, whether or not study treatment was received. The ITT population was analyzed according to the treatment assigned at randomization. Overall survival was assessed on participants randomized at least 15 days prior to the clinical cutoff date of December 30, 2010.
Measure: Number; unit: participants
Arm/Group | Vemurafenib | Dacarbazine
Number analyzed (Participants) | 336 | 336
participants
  Participants with events | 43 | 75
  Participants without events | 293 | 261
Statistical Analysis 1: Comparison: Vemurafenib vs Dacarbazine; The trial had a power of 80% to detect a hazard ratio of 0.65 for overall survival with an alpha level of 0.045 (an increase in median survival from 8 months for dacarbazine to 12.3 months for vemurafenib), one interim analysis for overall survival at 50% information; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.37, 95% CI 2-sided [0.26 to 0.55] — The hazard ratio for death for vemurafenib relative to dacarbazine and the associated 95% confidence interval were computed using an unstratified Cox regression model

2. Primary Outcome: Progression-free Survival
Description: A progression-free survival (PFS) event was defined as disease progression or death due to any cause. Tumor response (progression) was assessed according to the Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 criteria using computed tomography (CT) scans or magnetic resonance imaging (MRI).
Time Frame: From randomization (initiated January 2010) to December 30 2010.
Population: The analysis population for PFS consisted of all ITT participants randomized by October 27, 2010 (at least 9 weeks prior to the clinical cutoff date of December 30, 2010). The 9-week interval was chosen to allow time for participants to have had their first scheduled post baseline tumor assessment CT scan.
Measure: Number; unit: participants
Arm/Group | Vemurafenib | Dacarbazine
Number analyzed (Participants) | 275 | 274
participants
  Participants with events | 104 | 182
  Participants without events | 171 | 92
Statistical Analysis 1: Comparison: Vemurafenib vs Dacarbazine; The trial had a power of 90% to detect a hazard ratio of 0.55 for progression-free survival with an alpha level of 0.005 (an increase in median survival from 2.5 months for dacarbazine to 4.5 months for vemurafenib); Test type: Superiority or Other; p < .0001, Log Rank; Hazard Ratio (HR) = 0.26, 95% CI 2-sided [0.20 to 0.33] — Hazard ratios for treatment with vemurafenib, as compared with dacarbazine, were estimated with the use of unstratified Cox regression

3. Secondary Outcome: Participants With a Best Overall Response (BOR) of Complete Response or Partial Response
Description: BOR was defined as a complete response (CR) or partial response (PR) confirmed per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. Participants who never received study treatment and treated participants without any post-baseline tumor assessments were considered as non-responders. CR: Disappearance of all target lesions, all non-target lesions and no new lesion. Any pathological lymph nodes must have had reduction in the short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion and no new lesion.
Time Frame: From randomization (initiated January 2010) until December 30, 2010
Population: The analysis population consisted of all ITT participants randomized by September 22, 2010 (at least 14 weeks prior to the clinical cutoff date of December 30, 2010). The 14-week interval was chosen as it was the minimum time needed to observe a confirmed overall response according to protocol-specified schedule for the first two tumor assessments.
Measure: Number; unit: participants
Arm/Group | Vemurafenib | Dacarbazine
Number analyzed (Participants) | 219 | 220
participants
  Responders | 106 | 12
  Non-responders | 113 | 208

4. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time between the date of the earliest qualifying response and the date of disease progression or death due to any cause. Duration of response was calculated only for participants who had a best overall response of Complete Response or Partial Response and was estimated using the Kaplan-Meier method.
Time Frame: From randomization (initiated in January 2010) until December 30, 2010.
Population: The analysis population included all participants randomized by September 22, 2010 and with a best overall confirmed response of complete response or partial response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vemurafenib | Dacarbazine
Number analyzed (Participants) | 106 | 12
months | 5.49 [3.98 to 5.72] | NA [4.60 to NA] — Median duration of response was not reached as only 2 of the 12 participants with a qualifying response had subsequent disease progression or death due to any cause at the time of the analysis.

5. Secondary Outcome: Time to Confirmed Response
Description: Time to response was defined as the time from randomization to confirmed response (complete response or partial response).
Time Frame: From randomization (initiated January 2010) until December 30, 2010.
Population: as for outcome 4
Measure: Median (Full Range); unit: months
Arm/Group | Vemurafenib | Dacarbazine
Number analyzed (Participants) | 106 | 12
months | 1.45 [1.0 to 5.5] | 2.72 [1.6 to 5.8]

6. Secondary Outcome: Time to Treatment Failure
Description: Treatment failure was defined as a secondary endpoint in the protocol, defined as death, disease progression or premature withdrawal of study treatment. This endpoint was not included in the Statistical analysis plan; therefore no analyses of time to treatment failure were performed.
Time Frame: approximately 3 years
Arm/Group | Vemurafenib | Dacarbazine
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: The intensity of AEs was graded according to the NCI Common Terminology Criteria for Adverse Events v 4.0 (CTCAE) on a five-point scale (Grade 1 to 5: Mild, Moderate, Severe, Life-threatening and Death). A serious adverse event is any experience that suggests a significant hazard, contraindication, side effect or precaution, for example is life-threatening, requires hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or requires intervention to prevent one or other of the outcomes listed above.
Time Frame: From randomization (initiated January 2010) until December 30, 2010.
Population: The safety population was defined as all treated participants who had at least one on-study assessment. The safety population was analyzed according to the treatment received.
Measure: Number; unit: participants
Arm/Group | Vemurafenib | Dacarbazine
Number analyzed (Participants) | 336 | 282
participants
  Any adverse event | 326 | 253
  Serious adverse event | 110 | 45

8. Secondary Outcome: Pre and Post-dose Plasma Vemurafenib Concentration by Study Day
Description: The pharmacokinetics of vemurafenib were assessed at the beginning of each 21-day cycle using pre-dose and 2-4 hours post-dose sampling.
Time Frame: Plasma samples were collected before the morning dose (troughs) and 2-4 hours after the morning dose at the beginning of each cycle (Days 1, 22, 43, 64, 106, 148 and 190).
Population: The pharmacokinetic (PK) analysis population included all participants who received vemurafenib and provided valid PK assessments. The PK population at specific time points varied depending on the availability of confirmed dosing and PK assessment times. "n" indicates the number of participants with available PK data at each time point.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Vemurafenib
Number analyzed (Participants) | 260
μg/mL
  Pre-Dose Day 1 (n = 260) | 0 (0)
  Post-Dose Day 1 (n = 255) | 4.3 (4.35)
  Pre-Dose Day 22 (n = 204) | 53.0 (26.66)
  Post-Dose Day 22 (n = 221) | 54.0 (25.67)
  Pre-Dose Day 43 (n = 166) | 54.4 (24.13)
  Post-Dose Day 43 (n = 170) | 54.4 (23.28)
  Pre-Dose Day 64 (n = 141) | 57.4 (23.79)
  Post-Dose Day 64 (n = 138) | 57.7 (22.29)
  Pre-Dose Day 106 (n = 77) | 55.0 (17.62)
  Post-Dose Day 106 (n = 75) | 56.3 (20.36)
  Pre-Dose Day 148 (n = 38) | 51.8 (24.13)
  Post-Dose Day 148 (n = 39) | 53.3 (21.55)
  Pre-Dose Day 190 (n = 9) | 53.6 (12.6)
  Post-Dose Day 190 (n = 9) | 50.5 (20.16)

ADVERSE EVENTS:
Time Frame: Baseline through the end of study (maximum exposure: 57.07 months)
Groups:
- Vemurafenib: Adverse events reported for this group include those occurring in participants receiving vemurafenib starting at their baseline visit.
  Participants received continuous oral doses of vemurafenib (RO5185426) 960 mg twice a day. Participants took four 240 mg tablets in the morning and four 240 mg tablets in the evening (960 mg twice a day for a total daily dose of 1920 mg).
- Dacarbazine: Adverse events reported for this group include those occurring in participants receiving dacarbazine starting at their baseline visit until study discontinuation or treatment switch.
  Dacarbazine was administered intravenously 1000 mg/m˄2 up to 60 minutes on Day 1 of every 3 weeks (3 weeks was one cycle length).
- Vemurafenib After Crossover: Adverse events reported for this group include those occurring following switch to vemurafenib in those participants who switched from dacarbazine to vemurafenib during the study.
Arm/Group | Vemurafenib | Dacarbazine | Vemurafenib After Crossover
Serious Adverse Events (participants affected / at risk) | 165/336 | 52/293 | 44/84
Other Adverse Events (participants affected / at risk) | 333/336 | 247/293 | 83/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib (N=336) | Dacarbazine (N=293) | Vemurafenib After Crossover (N=84)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0
Orbital oedema (Eye disorders) | 1 | 0 | 0
Uveitis (Eye disorders) | 3 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 3 | 0 | 0
Device occlusion (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 2 | 1 | 1
Gait disturbance (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 5 | 4 | 3
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Encephalitis (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Herpes virus infection (Infections and infestations) | 1 | 0 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 2 | 2
Sepsis (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 2
International normalised ratio decreased (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 2 | 3
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 36 | 3 | 6
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 66 | 2 | 12
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 2 | 0 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 2 | 0 | 1
Sensorimotor disorder (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 1 | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Shock (Vascular disorders) | 0 | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 2 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib (N=336) | Dacarbazine (N=293) | Vemurafenib After Crossover (N=84)
Anaemia (Blood and lymphatic system disorders) | 32 | 22 | 13
Neutropenia (Blood and lymphatic system disorders) | 1 | 34 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 20 | 1
Abdominal Distension (Gastrointestinal disorders) | 18 | 5 | 2
Abdominal Pain (Gastrointestinal disorders) | 35 | 12 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 37 | 8 | 5
Constipation (Gastrointestinal disorders) | 52 | 72 | 8
Diarrhoea (Gastrointestinal disorders) | 124 | 36 | 24
Dyspepsia (Gastrointestinal disorders) | 20 | 2 | 2
Nausea (Gastrointestinal disorders) | 132 | 128 | 33
Vomiting (Gastrointestinal disorders) | 73 | 77 | 20
Asthenia (General disorders) | 50 | 29 | 7
Chest Pain (General disorders) | 26 | 5 | 4
Chills (General disorders) | 23 | 3 | 2
Fatigue (General disorders) | 158 | 101 | 32
Influenza Like Illness (General disorders) | 29 | 5 | 3
Oedema Peripheral (General disorders) | 49 | 15 | 8
Pain (General disorders) | 30 | 14 | 2
Peripheral Swelling (General disorders) | 26 | 0 | 5
Pyrexia (General disorders) | 71 | 26 | 18
Conjunctivitis (Infections and infestations) | 20 | 1 | 2
Folliculitis (Infections and infestations) | 28 | 3 | 2
Influenza (Infections and infestations) | 18 | 4 | 3
Nasopharyngitis (Infections and infestations) | 36 | 10 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 19 | 5 | 4
Sunburn (Injury, poisoning and procedural complications) | 57 | 0 | 15
Alanine Aminotransferase Increased (Investigations) | 28 | 4 | 6
Aspartate Aminotransferase Increased (Investigations) | 25 | 3 | 8
Blood Alkaline Phosphatase Increased (Investigations) | 33 | 0 | 9
Blood Bilirubin Increased (Investigations) | 31 | 1 | 2
Blood Creatinine Increased (Investigations) | 28 | 1 | 7
Gamma-Glutamyltransferase Increased (Investigations) | 24 | 4 | 7
Weight Decreased (Investigations) | 32 | 8 | 4
Decreased Appetite (Metabolism and nutrition disorders) | 76 | 24 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 189 | 9 | 48
Back Pain (Musculoskeletal and connective tissue disorders) | 53 | 20 | 11
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 44 | 11 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 50 | 5 | 15
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 76 | 18 | 14
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 39 | 3 | 9
Seborrhoeic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 46 | 2 | 8
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 96 | 1 | 17
Dizziness (Nervous system disorders) | 41 | 14 | 3
Dysgeusia (Nervous system disorders) | 55 | 10 | 9
Headache (Nervous system disorders) | 113 | 29 | 23
Hyperaesthesia (Nervous system disorders) | 17 | 1 | 0
Paraesthesia (Nervous system disorders) | 30 | 16 | 6
Depression (Psychiatric disorders) | 21 | 7 | 3
Insomnia (Psychiatric disorders) | 37 | 16 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 52 | 24 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33 | 24 | 8
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 27 | 5 | 3
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 44 | 12 | 13
Alopecia (Skin and subcutaneous tissue disorders) | 162 | 7 | 25
Dermal Cyst (Skin and subcutaneous tissue disorders) | 26 | 1 | 3
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 18 | 1 | 4
Dry Skin (Skin and subcutaneous tissue disorders) | 80 | 2 | 16
Erythema (Skin and subcutaneous tissue disorders) | 61 | 4 | 12
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 99 | 1 | 15
Keratosis Pilaris (Skin and subcutaneous tissue disorders) | 32 | 1 | 7
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 34 | 2 | 11
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 136 | 13 | 26
Pruritus (Skin and subcutaneous tissue disorders) | 86 | 5 | 14
Rash (Skin and subcutaneous tissue disorders) | 143 | 6 | 28
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 34 | 1 | 10
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 18 | 0 | 2
Skin Lesion (Skin and subcutaneous tissue disorders) | 40 | 4 | 4
Flushing (Vascular disorders) | 17 | 6 | 2
Lower respiratory tract infection (Infections and infestations) | 8 | 2 | 6
Urinary tract infection (Infections and infestations) | 9 | 9 | 5
Acne (Skin and subcutaneous tissue disorders) | 15 | 0 | 5
Rash erythematous (Skin and subcutaneous tissue disorders) | 9 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.